# 義大醫療財團法人義大醫院人體試驗委員會

# 臨床試驗受試者同意書

(送件時主持人請在此處

(本同意書應由計畫主持人親自向受試者說明詳細內容,並請受試者經過慎重考慮後万得簽名)

您被邀請參與此項研究,或您代理受試者同意被邀請參與此次研究,本表格提供您有關本研究的相關資訊。本項研究已通過本院人體試驗委會之審查通過 (人體試驗委員會編號: EMRP15107N)。計劃主持人將親自向您說明研究的詳細內容並回答

您的任何疑問,請經過慎重考慮後方予簽名。

(受試者編號: )

# 計畫名稱

中文:探討插管前給氧的氧氣分壓濃度對手術全期併發症之影響

英文: Effects of Preoxygenation with Lower Fraction of Inspired Oxygen during Induction of Anesthesia.

執行單位:義大醫療麻醉部

委託單位/藥廠:

主要主持人: 林真福 機構/職稱: 義大醫院/麻醉部部長 電話: 615-0011 轉 253045 共同主持人: 李匡曜 機構/職稱: 義大醫院/麻醉部主治醫師 電話: 615-0011 轉 253155 共同主持人: 蘇子桓 機構/職稱: 義大醫院/麻醉部住院醫師 電話: 615-0011 轉 252913 協同主持人: 蔡佩容 機構/職稱: 義大醫院/護理部高專 電話: 615-0011 轉 257063 協同主持人: 蔡依玲 機構/職稱: 癌治療醫院/麻醉專科護理師 電話: 615-0011 轉 257057 協同主持人: 蘇欣瑩 機構/職稱: 大昌醫院/麻醉專科護理師 電話: 615-0011 轉 258330

※二十四小時緊急聯絡人:蘇子桓 電話:0918-087-529

| 並 | ユよ | +2 | 1L | 27 | • |
|---|----|----|----|----|---|
| 攵 | 缸 | 石 | 姓 | 石 | • |

性別: 出生日期:

病歷號碼:

通訊地址:

聯絡電話:

法定代理人/有同意權人姓名:

與受試者關係:

性別: 出生日期:

身份證字號:

通訊地址:

聯絡電話:

版本: 第二版 日期: 2018 年 7 月 5 日 

#### 1.新醫療技術在全球執行情形或現況簡介:

臨床上常規使用純氧進行插管前給氧,以降低病人在進行全身麻醉誘導時低血氧發生之風險。然而這個作法並沒有臨床實證等級依據,尤其近來兩個大規模的臨床試驗結果,並不支持常規性給予急性心肌梗塞或是急性腦中風病人純氧氣補充,高濃度氧氣治療不僅對這類重大急症沒有治療上的效果,甚至可能顯著地增加治療患者的死亡率(血氧飽和濃度>94-96%)。另外,已有實驗證明高濃度氧氣對人體有害,特別是過氧化物的生成可能造成肺臟組織傷害,吸收性肺塌陷等相關併發症之發生率也可能增加。所以就目前臨床實證醫學來說,並沒有明顯證據可佐證麻醉前給予純氧有絕對好處,但高濃度氧氣治療所導致的傷害卻是越來越被廣泛關注的重要議題;換句話說,麻醉前給予較低濃度氧氣的風險相當低,而給予較高濃度氧氣反倒可能産生相當嚴重的術後併發症。

#### 2.試驗目的:

本試驗欲比較在沒有潛在低血氧風險的病人身上使用純氧或是較低氧氣分壓(FiO<sub>2</sub>=0.6)進行插管前給氧後,觀察在執行插管過程中低血氧之發生率及手術後七天內的併發症發生率是否有所差異,進而探討麻醉誘導期之給氧濃度對全身麻醉及手術後結果的影響。

3.試驗預計執行期間、受試驗者數目、收案地點/來源:

執行期間:自人體試驗委員會審核通過 起至西元 2019 年 12 月 31 日止

受試驗者數目:1000-1500 人

收案地點/來源:在義大醫院、義大癌治療醫院及義大大昌醫院接受氣管內插管全身麻醉 手術之病人

4.試驗之主要納入與排除條件:

<u>試驗者主要納入條件</u>: 1)您將在義大醫院、義大癌醫院或義大大昌醫院接受氣管內插管全身麻醉手術。2)您的年齡介於 20 到 65 歲之間。3)您屬於美國麻醉醫師協會麻醉風險等級 American Society of Anesthesiologists (ASA) I- III 的病人。

試驗者主要排除條件: 1)您有困難插管、困難換氣之風險。2)您患有嚴重的肺部疾病(包括急性上呼吸道感染)。3)您被診斷為冠狀動脈疾病或心肌梗塞。4)您患有嚴重的心衰竭疾病(NYHA Fc≥III)。5)您有肝功能異常或肝硬化,經臨床醫師評估為 Child-Pughs class B或 C。6)您患有急性或慢性腎病變(血清肌酸酐 Creatinine≥2 mg/dl)。7)您患有嚴重貧血(血紅素低於8 mg/dl)。8)您的 BMI>35。9)您目前已懷孕。10)您的空腹(禁食)時間不足,或是有腸阻塞、嚴重胃食道逆流等高吸入性肺炎風險。11)您接受的手術種類:緊急手術、開顱手術、心臟手術、肺部手術等。12)您為無行為能力、限制行為能力或意識不清、失智症、智能障礙等無法自主同意之病人。13)您拒絕參與此實驗計畫。

#### 5.試驗方法及相關檢驗:

- 1) 您符合納入條件且同意加入本研究計畫後,會以隨機分配的方式決定您的分組為高濃度氧氣(FiO2=1)組或是低濃度氧氣(FiO2=0.6)組。隨機分配由非執行臨床麻醉的臨床統計師按照事前已制定好的亂碼表指定您的治療組別。
- 2) 您在手術當天進入手術室後,會依常規放置血氧濃度計及其他生理監測計,隨後由訓練合格的麻醉科護理師或麻醉科醫師(包括住院醫師及主治醫師) 執行插管前給氧,並請您以每60秒8-10次之頻率進行自發性深呼吸。在您因麻醉誘導及肌肉鬆弛劑注射而失去自發性呼吸後,給予適當之正壓通氣直到進行插管動作。
- 3) 手術前後您的各項生理測量值將詳細記錄。
- 4) 本試驗無其他試驗用藥或是安慰劑使用,也沒有抽血等採集檢體之行為。
- 6.剩餘檢體處理情形:

此研究並沒有採用任何檢體。

### 7.可能產生之副作用、發生率及處理方法:

- 1.較低氧氣濃度治療組(FiO<sub>2</sub>= 0.6)可能發生麻醉誘導後低血氧現象。因為麻醉全程皆有相關生理監測系統進行血氧分析,而且有麻醉醫師及護理師隨時在場,任何低血氧的狀況皆會按照臨床標準作業執行處理,短時間的低血氧在適當的臨床處置後是不會有任何後遺症的。
- 2.處理方式:給予較高濃度氧氣、適當之正壓通氣、增加每分鐘通氣量,並持續監測血氧 濃度。

#### 8.其他替代療法及說明:

本試驗受試者與常規接受氣管內插管全身麻醉手術之病人,在處置上僅有插管前給氧之氧氣濃度不同,在密集生理監測及標準作業處理之下,不影響受試者的治療與預後。

#### 9. 試驗預期效益:

目前對於臨床麻醉中常規給予純氧作插管前給氧治療並無臨床實證支持,也尚未有研究 證實以較低氧氣分壓進行麻醉誘導給氧時,是否能減少手術全期可能由於氧氣毒性而產 生之肺損傷或細胞損傷。因此本臨床研究成果可提供在一般病人於麻醉插管前常規給氧 濃度之臨床實證依據,並確立麻醉誘導期之給氧濃度對全身麻醉及手術後結果的影響。

#### 10.試驗進行中受試者之禁忌、限制與應配合之事項:

- 1) 一切術前準備 (包含點滴給予、空腹禁食時間等)皆依常規進行。
- 2) 進行插管前給氧時,請病人配合以每 60 秒 8-10 次之頻率進行自發性深呼吸,與常規作法完全一致。

#### 11.機密性:

- A. 本研究依衛生福利部與本院人體試驗委員會之要求,妥善保存您的相關資料。
- B. 經由簽署受試者同意書,您瞭解亦同意研究贊助者、衛生福利部與本院人體試驗委員會皆有權檢視受試者的醫療記錄,以確保臨床研究過程與數據符合相關法律及法規要求。我們也承諾在法律所規範之程度內絕對視受試者的資料為機密並負有保密之義務。
- C. 有關辨認受試者身份之紀錄在相關法律及法規要求下不會予以公開。如果發表研究結果,受試者的身份仍將被保密。
- 12.補助、所需費用、損害賠償與保險:
- A. 參加試驗之補助:參加本研究,無任何補助。
- B. 費用負擔:參加本試驗您不需負擔任何與本試驗相關之費用或您應支付之費用。
- C. 如依本研究所訂臨床試驗計畫,因而發生不良反應或傷害,由<u>義大醫院</u>負損害補償責任。但本受試者同意書上所記載之可預期不良反應,不予補償。
- D. 如依本研究所訂試驗計畫,因而發生不良反應或損害,義大醫院願意提供專業醫療照 顧及醫療諮詢,您不必負擔治療不良反應或損害之必要醫療費用。
- E. 除前項賠償及醫療照顧外,本研究不提供其他形式之補償。若您不願意接受這樣的風險,請勿參加本研究計畫。
- F.您不會因為簽署本同意書或不簽署本同意書,而喪失在法律上的任何權利。

#### 13.受試者權利:

參加本研究計畫受試者個人權益將受到保護

- A. 研究過程中,與受試者的健康或疾病有關的任何發現,可能影響您繼續接受參與研究的意願,都將即時提供您。
- B. 如果您在研究過程中對研究工作性質產生疑問,對身為患者之權利有意見或懷疑因參 與研究而受害時,可與本院之人體試驗委員會聯絡請求諮詢,其電話號碼為 07-6151100


#### 轉分機 5110/5111。

- C. 如果您現在或於研究期間有任何問題或狀況,請隨時聯絡計劃共同主持人蘇子桓,其電話為:07-6150011轉分機 252913,手機 0918087529。
- D. 本同意書一式兩份,醫師已將同意書副本交給你(妳),並已完整說明本研究之性質與 目的。主持人<u>林真福</u>已回答您有關此研究相關的問題。
- 14.研究可能衍生之成果、商業利益與其應用之約定
- A. 如本院之研究計劃成果獲得學術文獻發表、智慧財產時,受試者同意無償供本院作為 從事疾病診斷、預防治療及研究醫學之用途。
- B. 本研究預期不會衍生專利權或其他商業利益。

#### 15.試驗之退出與中止:

您可自由決定是否參加本試驗;試驗過程中也可隨時撤銷同意,退出試驗,不需任何理由,且不會引起任何不愉快或影響其日後醫師對您的醫療照顧。試驗主持人亦可能於必要時中止該試驗之進行。

版本: 第二版 日期: 2018 年 7 月 5 日 

## 16.簽名:

- (一)受試者已詳細瞭解上述研究方法及其所可能產生的危險與利益,有關本試驗計畫的疑問,業經計畫主持人詳細予以解釋。本人同意接受為臨床試驗計畫的自願受試者。
- 1.受試者<u>為無行為能力</u>(未滿七歲之兒童<u>或受監護宣告之人</u>),應得其法定代理人或監護人之 同意。
- 2.限制行為能力人(滿七歲以上至未滿 20 歲或受輔助宣告之人),應得其本人及法定代理人或輔助人共同同意並簽署同意書。
- 3.<u>受試者雖非無行為能力或限制行為能力者,但無法自行簽署同意書時</u>,應由有同意權人為 之。(同意順序依相關法律規定辦理)。

| 受試者簽名: |
|---|
| 法定代理人/監護人/輔助人/有同意權人簽名(如適用): |
| 與受試者關係: 日期:西元 年 月 (二)見證人使用時機: 1.受試者、法定代理人或有同意權之人皆無法閱讀時,應由見證人在場參與所有有關受試者同意書之討論。見證人應閱讀受試者同意書及提供受試者之任何其他書面資料,以見證試驗主持人或其指定之人員已經確切地將其內容向受試者、法定代理人或有同意權之人解釋,並確定其充分了解所有資料之內容。 2.受試者、法定代理人或有同意權之人,仍應於受試者同意書親筆簽名並載明日期。但得以 |
| 與受試者關係: 日期:西元 年 月 (二)見證人使用時機: 1.受試者、法定代理人或有同意權之人皆無法閱讀時,應由見證人在場參與所有有關受試者同意書之討論。見證人應閱讀受試者同意書及提供受試者之任何其他書面資料,以見證試驗主持人或其指定之人員已經確切地將其內容向受試者、法定代理人或有同意權之人解釋,並確定其充分了解所有資料之內容。 2.受試者、法定代理人或有同意權之人,仍應於受試者同意書親筆簽名並載明日期。但得以 |
| 日期:西元 |
| <ul> <li>(二)見證人使用時機:</li> <li>1.受試者、法定代理人或有同意權之人皆無法閱讀時,應由見證人在場參與所有有關受試者同意書之討論。見證人應閱讀受試者同意書及提供受試者之任何其他書面資料,以見證試驗主持人或其指定之人員已經確切地將其內容向受試者、法定代理人或有同意權之人解釋,並確定其充分了解所有資料之內容。</li> <li>2.受試者、法定代理人或有同意權之人,仍應於受試者同意書親筆簽名並載明日期。但得以</li> </ul> |
| 1.受試者、法定代理人或有同意權之人皆無法閱讀時,應由見證人在場參與所有有關受試者<br>同意書之討論。見證人應閱讀受試者同意書及提供受試者之任何其他書面資料,以見證試<br>驗主持人或其指定之人員已經確切地將其內容向受試者、法定代理人或有同意權之人解<br>釋,並確定其充分了解所有資料之內容。<br>2.受試者、法定代理人或有同意權之人,仍應於受試者同意書親筆簽名並載明日期。但得以 |
| 同意書之討論。見證人應閱讀受試者同意書及提供受試者之任何其他書面資料,以見證試驗主持人或其指定之人員已經確切地將其內容向受試者、法定代理人或有同意權之人解釋,並確定其充分了解所有資料之內容。<br>2.受試者、法定代理人或有同意權之人,仍應於受試者同意書親筆簽名並載明日期。但得以 |
| 驗主持人或其指定之人員已經確切地將其內容向受試者、法定代理人或有同意權之人解釋,並確定其充分了解所有資料之內容。<br>2.受試者、法定代理人或有同意權之人,仍應於受試者同意書親筆簽名並載明日期。但得以 |
| 釋,並確定其充分了解所有資料之內容。<br>2.受試者、法定代理人或有同意權之人,仍應於受試者同意書親筆簽名並載明日期。但得以 |
| 2.受試者、法定代理人或有同意權之人,仍應於受試者同意書親筆簽名並載明日期。但得以 |
| 2.受試者、法定代理人或有同意權之人,仍應於受試者同意書親筆簽名並載明日期。但得以 |
| 3. 見證人於完成口述說明,並確定受試者、法定代理人或有同意權之人之同意完全出於其自 |
| 由意願後,應於受試者同意書簽名並載明日期。 |
| 4.試驗相關人員不得為見證人。 |
| 見證人簽名1:日期:西元年月日 |
| 見證人簽名 2:日期:西元 |

| 產生的危險與利益。 | | | | | |
|-----------------------|---------|----------|---|----|---|
| ● 取得受試者同意之人員 | (請打勾): | | | | |
| □ 研究人員/助理;簽名:_ | | _;日期:西元_ | £ | 年月 | 日 |
| □ 協同主持人 | | | | | |
| □ 共同主持人 | | | | | |
| □ 主要主持人 | | | | | |
| ● <u>主持人簽名</u> (請勾選類另 | 1) | | | | |
| □主要主持人 □共同主持人 | □協同主持人: | | | | |
| 簽名: | _;日期:西元 | 年 | 月 | | |

(三)主持人或研究人員已詳細解釋有關本研究計畫中上述研究方法的性質與目的,及可能

版本: 第二版 日期: 2018 年 7 月 5 日 